CLINICAL TRIAL: NCT00463840
Title: A Phase I/II Study of Chemoradiation With Oxaliplatin and 5FU for Locally Advanced Pancreatic Cancer
Brief Title: Chemoradiation With Oxaliplatin and Fluorouracil (5FU) for Locally Advanced Pancreatic Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to slow accrual
Sponsor: NYU Langone Health (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-64; H11640 (Other: NYU); Sanofi-Aventis 0x 03-030 (Other: Sanofi-Aventis)
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Results first posted 2012-05-01 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-10

CONDITIONS: Pancreatic Cancer
Keywords: Locally advanced pancreatic cancer; oxaliplatin; chemoradiation; 5FU
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin; Fluorouracil; Radiation; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxaliplatin+ 5FU+ radiation (RT) /surgery /FOLFOX 6 (Experimental): Concurrent chemoradiation before surgery and FOLFOX6 regimen after surgery
  Radiation (RT) 180cGy daily x 5 days/week x 5 weeks, then additional 540 cGy in 3 fractions over a half week to pancreatic portal;
  Combined with :
  5FU 200 mg/m^2 daily by continuous intravenous infusion (CIV) x 5 weeks and weekly Oxaliplatin 60 mg/m^2, IV for 5 weeks (in Phase I, 30, 40, 50, and 60 mg/m^2 Oxaliplatin were tested).
  Observation for 2 weeks to assess dose-limiting toxicity (DLT)/Response. Surgery if deemed resectable.
  Then modified FOLFOX 6 for 6 cycles (2 weeks/cycle):
  Day 1 hour 0: Oxaliplatin 85 mg/m^2 intravenously (IV) + Leucovorin 350 mg IV over 2 hours; hour 2: 5FU 400 mg/m^2 IV bolus followed by 2400 mg/m^2 IV over 46 hours.
  Interventions: Drug: Oxaliplatin; Drug: 5FU; Radiation: Radiation; Procedure: Surgery; Drug: FOLFOX 6

INTERVENTIONS:
Drug: Oxaliplatin
  Other Names: Oxaliplatin: Eloxatin
Drug: 5FU
  Other Names: 5-Fluorouracil
Radiation: Radiation
Procedure: Surgery
Drug: FOLFOX 6 — this is an established regimen of Oxaliplatin+infusional 5FU/Leucovorin

SUMMARY:
The intention of this trial is to determine the maximum tolerated of the treatment combination and to evaluate its safety and efficacy.

DETAILED DESCRIPTION:
Previous studies have demonstrated that neoadjuvant chemoradiation can lead to improved survival with a portion of patients proceeding to resection. This trial will incorporate a similar trial structure using newer agents in patients who present with locally advanced unresectable pancreatic cancer. Specifically oxaliplatin will be used owing to its greater activity in comparison to cisplatin and favorable therapeutic index in combination with radiation compared to gemcitabine.

In summary, the primary outcome measure of the phase I portion of the trial is to determine the maximum tolerated dose of this combination. Following the determination of this dose, the phase II portion of the trial will characterize the toxicity of this regimen as well as evaluate for long-term efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically documented pancreatic adenocarcinoma deemed unresectable due to local involvement of vessels or organs
* Patients with a clear clinical diagnosis of localized pancreatic cancer deemed unresectable, who have undergone at least 2 biopsies which were not diagnostic of adenocarcinoma, may be entered at the discretion of the principal investigator.
* No prior chemotherapy or abdominal radiation therapy.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Clinically measurable or evaluable disease.
* Life expectancy of at least 12 weeks.
* Adequate bone marrow reserve, granulocyte count >= 1500/uL, platelet count >= 100,000/uL, hemoglobin >= 9 g/dL.
* Adequate renal function with creatinine =< 1.5 times upper limit of normal (ULN)
* Adequate biliary function with bilirubin < 3.0 g/dL (including patients who have been bypassed or treated with percutaneous drainage), serum glutamic pyruvic transaminase (SGPT) (alanine transaminase) =< 2.5
* Age > 18 years
* Signed informed consent.
* No known allergy to one of the study drugs
* For female patient of childbearing potential, neither pregnant nor breastfeeding, and under active contraception
* No prior malignancy within last 5 years
* No central nervous system metastases
* No peripheral neuropathy > grade2
* No other serious concomitant illness

Exclusion Criteria:

* Active infection or uncontrolled infection
* Presence of metastatic disease.
* Inadequate organ function as discussed above.
* Pregnancy
* Serious concomitant systemic disorder.
* Use of any investigational agent within a month of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-06; Primary Completion 2010-07 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Ryan, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - Bellevue Hospital, New York, New York
  - NYU Cancer Institute, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 24 patients were enrolled to this Ph I/II study between June 2004 and December 2009 at New York University Medical Center.
Pre-assignment Details: The efficacy and toxicity data were based on both Ph I and II.
Groups:
- Oxaliplatin+ 5FU+ Radiation (RT) /Surgery /FOLFOX 6: Concurrent chemoradiation before surgery and FOLFOX6 regimen after surgery:
  Radiation (RT) 180cGy daily x 5 days/week x 5 weeks, then additional 540 cGy in 3 fractions over a half week to pancreatic portal;
  Combined with :
  5FU 200 mg/m^2 daily by continuous intravenous infusion (CIV) x 5 weeks and weekly Oxaliplatin 60 mg/m^2, IV for 5 weeks (in Phase I, 30, 40, 50, and 60 mg/m^2 Oxaliplatin were tested).
  Observation for 2 weeks to assess dose-limiting toxicity (DLT)/Response. Surgery if deemed resectable.
  Then modified FOLFOX 6 for 6 cycles (2 weeks/cycle):
  Day 1 hour 0: Oxaliplatin 85 mg/m^2 intravenously (IV) + Leucovorin 350 mg IV over 2 hours; hour 2: 5FU 400 mg/m^2 IV bolus followed by 2400 mg/m^2 IV over 46 hours.
Period: Overall Study
Arm/Group | Oxaliplatin+ 5FU+ Radiation (RT) /Surgery /FOLFOX 6
Started | 24
Completed | 12
Not Completed | 12
Not completed — Disease progression | 7
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Oxaliplatin+ 5FU+ Radiation (RT) /Surgery /FOLFOX 6
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 9
Age, Continuous [Median (Full Range); unit: years] | 63.7 [46 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Resectability After Chemoradiation
Description: This is the number of patients whose tumors are resectable after the combination treatment of 5FU, oxaliplatin, and radiation (RT).
Time Frame: 7.5 weeks
Population: Based on intent-to-treat population.
Measure: Number; unit: participants
Arm/Group | Oxaliplatin+ 5FU+ Radiation (RT) /Surgery /FOLFOX 6
Number analyzed (Participants) | 24
participants | 2

2. Secondary Outcome: Median Overall Survival
Description: This is the time at which 50% of patients are alive from the trial entry .
Time Frame: up to 10 years since the start of the study
Population: Secondary Measure was not reported. Contacted PI. No new Data available.
Arm/Group | Oxaliplatin+ 5FU+ Radiation (RT) /Surgery /FOLFOX 6
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 8 months
Description: treating period plus 30 days after the last protocol treatment
Arm/Group | Oxaliplatin+ 5FU+ Radiation (RT) /Surgery /FOLFOX 6
Serious Adverse Events (participants affected / at risk) | 11/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxaliplatin+ 5FU+ Radiation (RT) /Surgery /FOLFOX 6 (N=24)
Leukocytes (Total Wbc) (Blood and lymphatic system disorders) | 1
Anorexia (Gastrointestinal disorders) | 2
Ascites (Non-Malignant) (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 5
Diarrhea Patients Without Colostomy (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal-Other (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Infection With Unknown Anc (Infections and infestations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Dizziness/Lightheadedness (Nervous system disorders) | 1
Neuropathy - Motor (Nervous system disorders) | 1
Abdominal Pain Or Cramping (Gastrointestinal disorders) | 1
Pulmonary-Other (Respiratory, thoracic and mediastinal disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oxaliplatin+ 5FU+ Radiation (RT) /Surgery /FOLFOX 6 (N=24)
Hemoglobin (Blood and lymphatic system disorders) | 10
Leukocytes (Total Wbc) (Blood and lymphatic system disorders) | 17
Lymphopenia (Blood and lymphatic system disorders) | 21
Neutrophils/Granulocytes (Anc/Agc) (Blood and lymphatic system disorders) | 11
Platelets (Blood and lymphatic system disorders) | 17
Sinus Tachycardia (Cardiac disorders) | 4
Edema (Cardiac disorders) | 6
Hypotension (Cardiac disorders) | 2
Fatigue (Lethargy, Malaise, Asthenia) (General disorders) | 21
Fever (In The Absence Of Neutropenia, Where Neutropenia Is Defined As Agc<1.0 X 10e9/L) (General disorders) | 3
Rigors, Chills (General disorders) | 3
Weight Loss (General disorders) | 7
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 5
Dry Skin (Skin and subcutaneous tissue disorders) | 2
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 4
Anorexia (Gastrointestinal disorders) | 21
Ascites (Non-Malignant) (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 13
Dehydration (Gastrointestinal disorders) | 2
Diarrhea Patients Without Colostomy (Gastrointestinal disorders) | 15
Dyspepsia/Heartburn (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 3
Gastrointestinal-Other (Gastrointestinal disorders) | 3
Mucositis Due To Radiation (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 19
Stomatitis/Pharyngitis (Oral/Pharyngeal Mucositis) (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 13
Alkaline Phosphatase (Investigations) | 10
Hypoalbuminemia (Metabolism and nutrition disorders) | 16
Serum Glutamic Oxaloacetic Transaminase (Hepatobiliary disorders) | 7
Serum Glutamic Pyruvic Transaminase (Hepatobiliary disorders) | 5
Infection Without Neutropenia (Infections and infestations) | 3
Bicarbonate (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 11
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 12
Hypokalemia (Metabolism and nutrition disorders) | 10
Hyponatremia (Metabolism and nutrition disorders) | 12
Dizziness/Lightheadedness (Nervous system disorders) | 2
Insomnia (Nervous system disorders) | 2
Neuropathy - Motor (Nervous system disorders) | 2
Neuropathy-Sensory (Nervous system disorders) | 13
Cataract (Eye disorders) | 4
Abdominal Pain Or Cramping (Gastrointestinal disorders) | 2
Chest Pain (Non-Cardiac And Non-Pleuritic) (General disorders) | 2
Pain-Other (General disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Hiccoughs (Hiccups, Singultus) (Respiratory, thoracic and mediastinal disorders) | 2

LIMITATIONS AND CAVEATS:
This study did not reach its target accrual due to slow accrual. Small number of patients were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes